CLINICAL TRIAL: NCT02553915
Title: Omega-3 Fatty Acids for MDD With High Inflammation: A Personalized Approach
Brief Title: Omega-3 Fatty Acids for Major Depressive Disorder With High Inflammation: A Personalized Approach
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AT008857-01
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder; Overweight; Inflammation
Keywords: Omega-3; EPA; Depression; Overweight; Inflammation; Eicosapentaenoic acid
MeSH Terms: conditions — Depressive Disorder, Major; Overweight; Inflammation; Depression | interventions — Eicosapentaenoic Acid; Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: Study compared 3 dosing regimens of eicosapentaenoic acid (EPA), 1 g/day, 2 g/day, and 4 g/day versus an inactive placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All the above were blinded to the interventions. Placebo and EPA capsules had identical appearances.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Soybean oil placebo capsules, 4 capsules daily for 12 weeks
  Interventions: Other: Placebo
- EPA 1 g/day (Experimental): Eicosapentaenoic acid (EPA) 1000 mg capsules, 1 daily (plus 3 placebo capsules) for 12 weeks
  Interventions: Other: Placebo; Drug: EPA 1 g/day
- EPA 2 g/day (Experimental): Eicosapentaenoic acid (EPA) 1000 mg capsules, 2 daily (plus 2 placebo capsules) for 12 weeks
  Interventions: Other: Placebo; Drug: EPA 2 g/day
- EPA 4 g/day (Experimental): Eicosapentaenoic acid (EPA) 1000 mg capsules, 4 daily for 12 weeks
  Interventions: Drug: EPA 4 g/day

INTERVENTIONS:
Other: Placebo — Soybean oil placebo
  Arms: EPA 1 g/day; EPA 2 g/day; Placebo
Drug: EPA 1 g/day — Omega-3 fatty acid extracted from fish oil, 1 g/day
  Other Names: Eicosapentaenoic acid; omega-3 fatty acid
  Arms: EPA 1 g/day
Drug: EPA 2 g/day — Omega-3 fatty acid extracted from fish oil, 2 g/day
  Other Names: Eicosapentaenoic acid; omega-3 fatty acid
  Arms: EPA 2 g/day
Drug: EPA 4 g/day — Omega-3 fatty acid extracted from fish oil, 4 g/day
  Other Names: Eicosapentaenoic acid; omega-3 fatty acid
  Arms: EPA 4 g/day

SUMMARY:
This project aims to evaluate whether a dose-response relationship exists between dose of polyunsaturated fatty acids (PUFA), delivered as eicosapentaenoic acid (EPA), and change in markers of inflammation, and whether these effects differ from placebo. A key secondary aim is to evaluate the antidepressant effectiveness of EPA in overweight adult outpatients with current major depressive disorder (MDD). To address these aims, the project will use a four-arm, randomized, parallel-group, placebo-controlled design comparing placebo versus three doses of EPA (1 gm/day, 2 gm/day, or 4 gm/day) administered over 12 weeks. The study is to be conducted at two sites: Emory University School of Medicine, and Massachusetts General Hospital. Eligible participants will be between the ages of 18-80 who have current MDD, are overweight, and who demonstrate peripheral inflammation, defined as an high sensitivity C-reactive protein (hs-CRP) level ≥ 3 mg/L. The primary outcome will be change in plasma interleukin-6 (IL-6) levels and/or mitogen-stimulated peripheral blood mononuclear cells (PBMC) Tumor Necrosis Factor-alpha (TNF-α) expression levels in EPA- versus placebo-treated participants. The results of this investigation are intended to be used to design and power a larger definitive test of the efficacy and biological effects of EPA in patients with major depressive disorder.

DETAILED DESCRIPTION:
This study will evaluate the anti-inflammatory effects and antidepressant efficacy and tolerability of EPA versus placebo in the treatment of MDD. The study design is a randomized, placebo-controlled, double-blind parallel-group dose-finding 12 week outpatient clinical trial. The study population will consist of outpatients who are overweight and suffer from MDD, who also demonstrate systemic inflammation. Three doses of EPA (1 gm/d, 2 gm/d, and 4 gm/d) will be compared against placebo. The study will be conducted at two sites: Emory University School of Medicine and Massachusetts General Hospital. The study will be conducted under the Food and Drug Administration Investigational New Drug (IND) 074150.

One hundred adult MDD patients (ages 18-80) will be randomized to enter the 12-week double-blind treatment period. Each of the four study arms (3 EPA arms and one placebo arm) will have 25 patients, with the expectation of 20 completers per arm, based on a 20% early termination rate. The subjects will be recruited through advertisements and clinical referrals from psychiatrists and general physicians who are treating overweight outpatients with MDD. Participants must agree not to significantly modify their diet during the 12 weeks of the study.

Due to the need for participants to have a hs-CRP ≥ 3 mg/L to be eligible for the study, two screening visits will be used to minimize expenses associated with screening. The screening period may extend up to 28 days prior to the baseline visit (Visit 3) if necessary to allow for time need for participant scheduling and allow for any required repeat laboratory testing.

Patients screened for the study and found to be eligible will return for their baseline visit after one week, during which no psychotropic medication or PUFAs will be administered. Patients must have an Inventory of Depressive Symptoms, Clinician rated (IDS-C30) total score ≥ 25 at the baseline visit in order to be eligible for randomization.

Patients will be randomized to one of four treatment arms: 1) EPA 1 mg/day; 2) EPA 2 mg/day; 3) EPA 4 mg/day; or 4) Placebo. Randomization will be in blocks of 4 with separate randomization schedules for each site.

Study materials will include:

1. Study capsules containing EPA-enriched omega-3, 1000 mg tabs, supplied by Nordic Naturals.
2. Placebo capsules matching the EPA 1000 mg tabs, also to be supplied by Nordic Naturals.

Documentation of the presence of any side-effect or adverse event (AE) will be completed by one of the treating psychiatrists at every visit by recording all spontaneously reported AEs, which will be classified as either mild, moderate, or severe. Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) terms. Patients shall be allowed to contact the investigator or a member of his staff at any time between visits concerning adverse events or worsening of symptoms.

All concomitant medications taken during the study will be recorded in the case report form, along with dosage information and start and stop dates. Drugs that may be taken by the patient include any prescription or over-the-counter medication not specifically excluded by the protocol. Patients requiring excluded drugs (including antidepressants, benzodiazepines, antipsychotics, psychostimulants, and mood stabilizing agents) will be discontinued from the study.

Patients may choose to withdraw from the study at any time.

Participants may be withdrawn by the investigator should any of the following occur:

1. severe, persistent intolerance to study medication
2. worsening of depressive symptoms such that the subject's safety is endangered (e.g. suicidality)
3. development of mania or psychotic symptoms
4. a serious adverse event (SAE) that is either: i) considered by the investigator to be possibly, probably, or definitely related to the study medication, or ii) places the subject at increased risk of harm if she were to continue in the study
5. persistent non-adherence to the study medication, defined as not taking between 80-120% of the study medication pills for two consecutive visits
6. development of pregnancy

Patients with MDD may experience worsening of their depression and/or the emergence of suicidal ideation and behavior (suicidality), whether or not they are taking antidepressant medications, and this risk may persist until MDD remission occurs. This guidance is consistent with global class labelling for antidepressants. Although there has been a long-standing concern that antidepressants may have a role in inducing worsening of depression and the emergence of suicidality in certain subjects, a causal role for antidepressants in inducing such behaviors has not been established. Nevertheless, subjects being treated with study medication will be observed closely for clinical worsening and suicidality, especially at the beginning and end of the course of treatment, or at the time of dose changes, either increases or decreases. Consideration will be given to possibly discontinuing the investigational product in subjects whose depression is persistently worse or whose emergent suicidality is severe or abrupt in onset or was not part of the subject's presenting symptoms. To assess suicidal ideation and behaviors, the CSSRS will be used in this trial.

The following symptoms, anxiety, agitation, panic attacks, insomnia, irritability, hostility, impulsivity, akathisia (psychomotor restlessness), hypomania, and mania, have been reported in patients being treated with antidepressants for MDD. Consideration will be given to possibly discontinuing the study medication in subjects for whom such symptoms are severe, abrupt in onset, or were not part of the subject's presenting symptoms.

Research participants are exited from the study should any of the following occur:

* Any emergent Columbia Suicide Severity Rating Scale (CSSRS) defined suicidal behavior
* A suicidal ideation score of 5 (indicating active suicidal ideation with specific plan and some level of intent) on the CSSRS
* In the absence of a CSSRS suicidal ideation score of 5 or CSSRS-defined suicidal behavior, the investigator determines the patient to have a significant short-term risk for a suicide attempt.

Any participant who becomes pregnant during the study will be withdrawn from the study. The investigator will collect pregnancy information, record it on the Pregnancy Form, and submit it to the lead site PI, Mark Rapaport, MD, via email within 2 weeks of learning of a participant's pregnancy. The participant will also be followed to determine the outcome of the pregnancy. Follow-up is expected to end approximately 8 weeks following the estimated delivery date. Any premature termination of the pregnancy will be reported. While pregnancy itself is not considered to be an adverse event (AE) or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE. A spontaneous abortion is always considered an SAE and will be reported as such.

All randomized participants who terminate the trial prior to the Week 12 visit will be asked to return for an early termination visit. The study team should complete all the Week 12 assessments at the study termination visit. All subjects who complete the trial or discontinue because of lack of response or side effects will receive treatment as clinically appropriate and will then be referred for appropriate follow-up care.

Blood will be collected and analyzed for the screening tests and biomarker analyses. Urine samples will be collected and analyzed with a toxicology screen and urinalysis. We will collect physical records in the form of questionnaires, phone screenings, and psychiatric interviews. We will request access to participants' medical records only for reasons related to patient safety. Participant case report forms will be kept in locked file cabinets in the offices of each study site.

Biological specimens are linked to the individual patient only through a unique research code. All documents that directly reveal the participant's identity, such as signed consent forms, are stored in charts that are marked on the outside only with the participant's code number.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Men or women aged 18-80 years.
* A primary psychiatric diagnosis of major depressive disorder (MDD), by Diagnostic and Statistical Manual-5th ed (DSM-5) using the Mini International Neuropsychiatric Interview (MINI v.7.0).
* A Screening and Baseline visit Inventory of Depressive Symptoms, Clinician rated (IDS-C30) total score ≥ 25.
* Currently overweight at screening, defined as BMI > 25 kg/m2.
* Screening visit high-sensitivity C-reactive protein concentration ≥ 3 mg/L.
* Willing to not significantly modify their diet from the time they sign consent through the end of study participation.

Exclusion Criteria:

* Use of any psychotropic agents within 2 weeks of baseline or at any time during the study, with the exception of prescription hypnotics (eszopiclone, zaleplon, zolpidem, suvorexant, ramelteon), diphenhydramine, or a stable daily dose of a benzodiazepine.
* Breastfeeding or pregnant women, women intending to become pregnant within 6 months of the screening visit, or women of child bearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, intrauterine device (IUD), status-post tubal ligation, or partner with vasectomy)
* Patients who, in the investigator's judgement, pose a current, serious suicidal or homicidal risk.
* Serious or unstable medical illness that in the investigator's opinion could compromise response to treatment or interpretation of study results.
* History of seizure disorder, except for childhood febrile seizures.
* Meeting DSM-5 criteria at any point in their lifetime, for any of the following: Neurocognitive Disorder, Psychotic Disorder, Bipolar disorder, Anorexia Nervosa
* Meeting DSM-5 criteria in the 3 months prior to the screening visit for any Substance Use Disorder (except nicotine or caffeine).
* Meeting DSM-5 criteria at screening for current obsessive compulsive disorder or bulimia nervosa.
* Presence of psychotic features at any time during the current major depressive episode.
* Any conditions or medications (within 1 week of baseline or during the trial) that might confound the biomarker findings, including: Regular ingestion of NSAIDs or Cyclooxygenase-2 (COX-2) inhibitors, or any use of oral steroids, immunosuppressants, interferon, chemotherapy, or anticoagulants (Patients will be instructed not to take a nonsteroidal antiinflammatory drug (NSAID) or COX-2 inhibitor in the 24 hours prior to a biomarker assessment visit), Malignancy not in remission for at least 1 year, Active autoimmune disorder or inflammatory bowel disease, Insulin-dependent diabetes mellitus.
* History of allergy to PUFA supplements.
* Laboratory evidence of undiagnosed hypothyroidism or change in treatment for hypothyroidism in the 3 months prior to screening.
* Patients who have failed to respond during the course of their current major depressive episode to >4 adequate antidepressant trials, defined as six weeks or more of treatment with the FDA-defined minimally effective dose.
* Patients who have taken a supplement of at least 1 g/day of omega 3 fatty acids for at least 6 weeks during the current major depressive episode.
* Patients who have had electroconvulsive therapy (ECT) during the current depressive episode or within 6 months of the screening visit.
* Patients who have taken supplements with omega-3 fatty acids (see Appendix A for list of products) within sixty (60) days of the screening visit.
* Patients who, at baseline, are consuming a diet that contains more than 3g/day of omega-3 FA, or who consume more than 3 meals of fatty fish per week.
* Patients who have a history of a bleeding disorder.
* Patients who have participated in another clinical trial of an investigational medication within 1 month of the screening visit.
* Patients who are currently in psychotherapy that was initiated within 90 days prior to the study screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Depression Clinical and Research Program at Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mischoulon D, Nierenberg AA, Schettler PJ, Kinkead BL, Fehling K, Martinson MA, Hyman Rapaport M. A double-blind, randomized controlled clinical trial comparing eicosapentaenoic acid versus docosahexaenoic acid for depression. J Clin Psychiatry. 2015 Jan;76(1):54-61. doi: 10.4088/JCP.14m08986. PMID 25272149
- [Result] Rapaport MH, Nierenberg AA, Schettler PJ, Kinkead B, Cardoos A, Walker R, Mischoulon D. Inflammation as a predictive biomarker for response to omega-3 fatty acids in major depressive disorder: a proof-of-concept study. Mol Psychiatry. 2016 Jan;21(1):71-9. doi: 10.1038/mp.2015.22. Epub 2015 Mar 24. PMID 25802980
- [Derived] Mischoulon D, Dunlop BW, Kinkead B, Schettler PJ, Lamon-Fava S, Rakofsky JJ, Nierenberg AA, Clain AJ, Mletzko Crowe T, Wong A, Felger JC, Sangermano L, Ziegler TR, Cusin C, Fisher LB, Fava M, Rapaport MH. Omega-3 Fatty Acids for Major Depressive Disorder With High Inflammation: A Randomized Dose-Finding Clinical Trial. J Clin Psychiatry. 2022 Aug 22;83(5):21m14074. doi: 10.4088/JCP.21m14074. PMID 36005883
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Started | 15 | 15 | 15 | 16
Completed | 11 | 14 | 12 | 13
Not Completed | 4 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Adults with major depressive disorder, overweight, with elevated hsCRP at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 14 | 13 | 13 | 16 | 56
  >=65 years | 1 | 2 | 1 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 42 (15) | 44 (15) | 46 (13) | 46 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 11 | 46
  Male | 3 | 4 | 3 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 7 | 2 | 5 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 7 | 12 | 9 | 6 | 34
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown / Not Reported | 1 | 1 | 0 | 1 | 3
  Hispanic or Latino | 3 | 1 | 3 | 1 | 8
  Not Hispanic or Latino | 12 | 14 | 12 | 15 | 53
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 16 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Plasma Concentration of Inflammatory Biomarkers IL-6 (pg/mL) and PBMC TNF-α (pg/mL)
Description: To evaluate whether a dose-response relationship exists between dose of EPA and decrease either in plasma interleukin-6 (IL-6) levels (pg/mL) or in mitogen-stimulated peripheral blood mononuclear cell (PBMC) Tumor Necrosis Factor-α (TNF-α) expression and secretion (pg/mL), when compared with placebo. Levels of inflammatory biomarkers were assessed at baseline (week 0) and at week 12 for comparison. Percent changes were calculated as relative to baseline values. Greater percent decrease indicates better outcome.
Time Frame: 12 weeks
Population: Study completers with available biomarker data
Measure: Mean (Standard Deviation); unit: percentage of change in plasma levels
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Number analyzed (Participants) | 10 | 13 | 11 | 13
percentage of change in plasma levels
  % Change in Plasma IL-6 (pg/mL) at 12 weeks | 1.92 (30.24) | -1.27 (28.37) | 7.19 (32.24) | 4.45 (40.16)
  % Change in PBMC TNF-alpha (pg/mL) at 12 weeks | 8.59 (45.82) | -0.19 (39.63) | 10.38 (80.36) | 28.54 (56.97)
Statistical Analysis 1: Comparison: Placebo vs EPA 1 g/Day vs EPA 2 g/Day vs EPA 4 g/Day; To evaluate whether a dose-response relationship exists between dose of EPA and decrease either in plasma IL-6 levels or in mitogen-stimulated PBMC TNF-α expression and secretion, when compared with placebo. [Time Frame: 12 weeks]. Comparisons were made within each arm pre and post 12 weeks of treatment; Test type: Other — Comparisons were made for each biomarker within each arm pre and post 12 weeks of treatment; p < 0.10, Kruskal-Wallis

2. Primary Outcome: Mean Change in Depression Severity Score (IDS-C30) After 12 Weeks of Treatment
Description: To evaluate whether EPA treatment produces a decrease in ratings of depression severity after 12 weeks of treatment, when compared with placebo-treated subjects. Comparison is made between pre-treatment and post-12 weeks treatment. Inventory of Depressive Symptomatology-30 item-Clinician Rated (IDS-C30) is a depression severity scale, where lower scores indicate less depressive severity and higher scores indicate greater severity. Minimum score is 0 (zero) and maximum score is 84.
Time Frame: 12 weeks
Population: Study completers with available IDS-C30 data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Number analyzed (Participants) | 10 | 14 | 11 | 13
score on a scale
  Baseline IDS-C30 Score | 36.6 (10.54) | 36.14 (7.15) | 31.36 (7.12) | 31.92 (5.44)
  Raw change at week 12 | -17.6 (7.82) | -12.07 (11.29) | -12.73 (17.32) | -16.15 (10.49)
Statistical Analysis 1: Comparison: Placebo vs EPA 1 g/Day vs EPA 2 g/Day vs EPA 4 g/Day; To evaluate: 1. whether EPA treatment produces a decrease in ratings of depression severity, when compared with placebo-treated subjects; and 2. whether the changes in IL-6 or mitogen- stimulated PBMC TNF-α expression mediate changes observed in ratings of depression. [Time Frame: 12 weeks]; Test type: Superiority; p < 0.1, ANOVA

3. Primary Outcome: Percent Change in IDS-C Score After 12 Weeks of Treatment
Description: To evaluate whether EPA treatment produces a decrease in ratings of depression severity, when compared with placebo-treated subjects; and whether the changes in IL-6 or mitogen- stimulated PBMC TNF-α expression will mediate changes observed in ratings of depression.
  Inventory of Depressive Symptomatology-30 item-Clinician Rated (IDS-C30) is a depression severity scale, where lower scores indicate less depressive severity and higher scores indicate greater severity. Minimum score is 0 (zero) and maximum score is 84. Change in score over 12 weeks (from week 0 to week12) is calculated as a percent change from baseline. Greater percent change in the negative direction indicates better outcome.
Time Frame: 12 weeks
Population: Study completers with available data
Measure: Mean (Standard Deviation); unit: percentage change in score
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Number analyzed (Participants) | 10 | 14 | 11 | 13
percentage change in score | -50.73 (25.24) | -34.52 (31.51) | -37.53 (50.92) | -51.4 (30.23)
Statistical Analysis 1: Comparison: Placebo vs EPA 1 g/Day vs EPA 2 g/Day vs EPA 4 g/Day; Change in IDS-C30 scores were compared pre and post 12 weeks of treatment with each intervention, within each arm; Test type: Other; p < 0.01, Kruskal-Wallis

4. Secondary Outcome: Percent Change in Plasma Concentrations of Mitogen-stimulated PBMC IL-6 (pg/mL) and Plasma Tumor Necrosis Factor (TNF)-α (pg/mL)
Description: To evaluate whether EPA treatment produces decreases in plasma levels of mitogen-stimulated PBMC IL-6 and TNF-α (both in in pg/mL). Percent change calculated by comparing week 12 to week 0 (baseline). Greater decrease (change in negative direction) indicates better outcome.
Time Frame: 12 weeks
Population: Study completers with available biomarker data
Measure: Mean (Standard Deviation); unit: percentage of change in plasma levels
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Number analyzed (Participants) | 10 | 14 | 11 | 13
percentage of change in plasma levels
  % Change in Plasma PBMC IL-6 (pg/mL) at 12 weeks | 41.6 (78.1) | -0.51 (67.93) | 101.48 (296.86) | 17.37 (65.73)
  % Change in Plasma TNF-α (pg/mL) at 12 weeks | 9.98 (27.99) | 0.22 (23.33) | -1.95 (18.63) | -10.13 (13.98)
Statistical Analysis 1: Comparison: Placebo vs EPA 1 g/Day vs EPA 2 g/Day vs EPA 4 g/Day; To evaluate whether EPA treatment produces decreases in mitogen-stimulated PBMC IL-6. [Time Frame: 12 weeks] Comparisons were made between pre and post treatment levels in each of the 4 treatment arms; Test type: Other — Exploratory; p < 0.1, Spearman Rank Order Correlation

5. Secondary Outcome: Percent Changes in Levels of Expression of Inflammation-related Genes for Interleukin (IL)-6 and Tumor Necrosis Factor (TNF)-α (in ΔΔCt Units)
Description: To evaluate whether EPA treatment produces decreases in the expression of inflammation pathway-related genes for IL-6 and TNF-α (in ΔΔCt units). Levels compared at week 0 (baseline) and at week 12 to obtain percent change from baseline. Greater decrease (change in negative direction) indicates better outcome.
Time Frame: 12 weeks
Population: Completers with available genetic marker data
Measure: Mean (Standard Deviation); unit: percentage of gene expression level
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Number analyzed (Participants) | 9 | 12 | 11 | 10
percentage of gene expression level
  % Change in IL-6 Gene expression (ΔΔCt) at 12 week | 109.22 (285.65) | 1426 (4573) | 16.03 (141.26) | 20.2 (172.23)
  % change in TNF-α Gene expression (ΔΔCt) at 12 wks | 93.56 (316.02) | 217.46 (692.42) | -36.09 (37.32) | -2.27 (58.24)
Statistical Analysis 1: Comparison: Placebo vs EPA 1 g/Day vs EPA 2 g/Day vs EPA 4 g/Day; To evaluate whether EPA treatment produces decreases in the expression of inflammation pathway-related genes. [Time Frame: 12 weeks] (We evaluated gene expression of IL-6 and TNF-α.); Test type: Other — Exploratory; p < 0.1, Spearman Rank Order Correlation

6. Secondary Outcome: Percent Change in High-sensitivity C-reactive Protein (Hs-CRP) in mg/L
Description: To evaluate whether EPA treatment produces decreases in plasma hs-CRP in mg/L. Levels compared at week o (baseline) and week 12 to obtain percent change. Greater percent decrease in the negative direction indicates better outcome.
Time Frame: 12 weeks
Population: Study completers with available biomarker data
Measure: Mean (Standard Deviation); unit: percentage of change in plasma levels
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
Number analyzed (Participants) | 10 | 13 | 11 | 13
percentage of change in plasma levels | 7.22 (54.27) | -9.52 (53.87) | 1.09 (74.46) | -17.96 (35.08)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded only if they emerged or worsened during the course of the study. Each patient was treated in the double blind protocol for 12 weeks. During this time, adverse events were inquired about and recorded as endorsed by patients.
Arm/Group | Placebo | EPA 1 g/Day | EPA 2 g/Day | EPA 4 g/Day
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 11/15 | 8/15 | 8/15 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | EPA 1 g/Day (N=15) | EPA 2 g/Day (N=15) | EPA 4 g/Day (N=16)
Abnormal Propulsive movement of large bowel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation alternating with diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea/Loose stool (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric reflux (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased frequency of bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Increased Urination (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Increased thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy symptoms (environmental) (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burn injury (right thumb) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst exacerbation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness of unknown cause (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (toe) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lower limb numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand laceration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tiredness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hives (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 4 (4)
Weight loss (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Smaller than projected sample due to challenges in recruitment led to smaller analyzable treatment arms. Results should be considered preliminary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT02553915/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT02553915/ICF_001.pdf